CLINICAL TRIAL: NCT03356132
Title: Post-market Monitoring and Control of Safety and Efficacy of Silimed® Breast Implants with Textured Surface and Polyurethane Foam-coated Surface
Brief Title: An Analysis of Adverse Events and Satisfaction Outcomes of Women Who Underwent Primary and Secondary Breast Augmentation Using Silimed® Breast Implants
Acronym: STEPS A
Status: Recruiting | Type: Observational
Sponsor: Silimed Industria de Implantes Ltda (Industry)
Responsible Party: Sponsor
Other Study IDs: 6002030
Record Dates: First submitted 2017-11-14; First posted 2017-11-29 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Breast Implant; Complications; Quality of Life; Satisfaction
Keywords: breast implant; complication; satisfaction; quality of life; augmentation; textured; polyurethane
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Textured Group: Women undergoing primary and secondary breast augmentation with Silimed® Textured Silicone Gel-Filled Breast Implant.
  Interventions: Device: Silimed® Textured Silicone Gel-Filled Breast Implant
- Polyurethane Group: Women undergoing primary and secondary breast augmentation with Silimed® Polyurethane Foam Covered Silicone Gel-Filled Breast Implant
  Interventions: Device: Silimed® Polyurethane Foam Covered Silicone Gel-Filled Breast Implant

INTERVENTIONS:
Device: Silimed® Textured Silicone Gel-Filled Breast Implant — Women undergoing primary and secondary breast augmentation using Silimed® Textured Silicone Gel-Filled Breast Implant.
  Groups: Textured Group
Device: Silimed® Polyurethane Foam Covered Silicone Gel-Filled Breast Implant — Women undergoing primary and secondary breast augmentation using Silimed® silicone gel-filled breast implants with polyurethane foam covered surface.
  Groups: Polyurethane Group

SUMMARY:
The study investigates the safety and performance of Silimed® silicone gel breast implants with a textured surface and Silimed® silicone gel breast implants with polyurethane coated surface. Female patients who underwent primary or secondary breast augmentation using Silimed® breast implants will be followed-up through 10 years. The safety of each type of Silimed® breast implant is going to be assessed by estimating the known and unexpected short- and long-term risk / adverse event rates. The performance of each type of Silimed® breast implant is going to be assesses by estimating the satisfaction and quality of life after implantation.

ELIGIBILITY:
Inclusion Criteria:

* provide written informed consent.
* female at birth
* be 18 years of age or older
* have received breast implant(s) for indication of primary or secondary augmentation until 21 days before (including the visit window)
* having received a breast implant with a textured surface or a breast implant with a surface coated with Silimed® polyurethane foam
* ability to comply with the protocol throughout the follow-up period.

Exclusion Criteria:

* mammary reconstruction in at least one breast or augmentation after previous reconstruction,
* pregnancy informed or breastfeeding at the inclusion moment,
* advanced fibrocystic disease at the time of implantation,
* neoplasia of any type not yet treated or being treated at the time of implantation, infection in activity not yet treated or being treated at any site at the time of implantation,
* reporting or recording of adverse reactions or intolerance to polyurethane or silicone prior to implantation,
* immune diseases affecting active connective tissue or (eg, lupus erythematosus, discoid lupus, scleroderma, etc.) at the time of implantation,
* signs of inflammation of the breast or implant site at the time of implantation,
* Increased risk of immediate postoperative complications due to use of illicit drugs or medications,
* Increased risk of immediate post-surgical complications caused by illicit drug use or medication use,
* have participated in another clinical study up to 6 months prior to the placement of the implant,
* any other condition which, based on the opinion of the investigator or designee, may prevent the provision of informed consent, renders participation in the study is unsafe, compromises adherence to the protocol, complicates the interpretation of data from the study outcome, or otherwise interferes with the achievement of study objectives.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women aged 18 years old or older who have undergone breast augmentation using Silimed® silicone gel-filled breast implants with textured surface or Silimed® silicone gel-filled breast implants with polyurethane foam coated surface.
Sampling Method: Non-Probability Sample
Enrollment: 632 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Expected Adverse Events | Every three years through the 10 years length of the study.
  Estimate the known short-term and long-term risk / adverse event rate for Silimed® silicone gel-filled breast implants with textured surface and Silimed® silicone gel-filled breast implants with polyurethane foam covered surface
Unexpected Adverse Events | Every three years through the 10 years length of the study.
  Estimate the unknown short-term and long-term risk / adverse event rate for Silimed® silicone gel-filled breast implants with textured surface and Silimed® silicone gel-filled breast implants with polyurethane foam covered surface

SECONDARY OUTCOMES:
Patient's Satisfaction in Relation to Aesthetic Result | Every three years through the 10 years length of the study.
  Estimate the performance of Silimed® silicone gel-filled breast implants with textured surface and Silimed® silicone gel-filled breast implants with polyurethane foam covered surface through the satisfaction of the patient regarding the aesthetic result after breast augmentation. The assessment of patient's satisfaction will be done by means of a likert scale, where the following satisfaction options can be selected: 1 = definitely satisfied, 2 = satisfied, 3 = slightly satisfied, 4 = slightly dissatisfied and 5 = definitely unsatisfied.
Patient's Satisfaction in General | Every three years through the 10 years length of the study.
  Estimate the performance of Silimed® silicone gel-filled breast implants with textured surface and Silimed® silicone gel-filled breast implants with polyurethane foam covered surface after breast augmentation by means of a questionnaire, the Breast Self-Assessment Questionnaire (BEQ-Brazil), which consist of 55 questions related to satisfaction and comfort with the overall appearance of the breasts.
Evaluator's Satisfaction in Relation to Aesthetic Result | Every three years through the 10 years length of the study.
  Estimate the performance of Silimed® silicone gel-filled breast implants with textured surface and Silimed® silicone gel-filled breast implants with polyurethane foam covered surface through the satisfaction of the evaluator regarding the aesthetic result after patient's breast augmentation. The assessment of evaluator's satisfaction will be done by means of a likert scale, where the following satisfaction options can be selected: 1 = definitely satisfied, 2 = satisfied, 3 = slightly satisfied, 4 = slightly dissatisfied and 5 = definitely unsatisfied.
Patient's Quality of Life | Every three years through the 10 years length of the study.
  Estimate the performance of Silimed® silicone gel-filled breast implants with textured surface and Silimed® silicone gel-filled breast implants with polyurethane foam covered surface through the quality of life of the patient after breast augmentation. The assessment of patient's quality of life will be done by means of the Rosemberg Global Self-Esteem Scale, in order to evaluate the overall self-esteem of the sample.

CONTACTS AND LOCATIONS:
Overall Officials: Celso EJ Boechat, MD, Principal Investigator — Perfektua Serviços Médicos Ltda
Locations (1):
- Perfektua Serviços Médicos Ltda, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The IPD will be shared starting 6 months after the end of the study.
Access Criteria: It was not defined yet.